CLINICAL TRIAL: NCT05364983
Title: A Prospective, Randomized, Controlled, Double-Masked, Phased, Multi-Center Clinical Study to Evaluate the Safety and Efficacy of the LensGen® Juvene® Intraocular Lens
Brief Title: Clinical Study to Evaluate the LensGen® Juvene® Intraocular Lens
Acronym: Nirvana
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LensGen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CP20-001
Record Dates: First submitted 2022-05-04; First posted 2022-05-06 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2022-05

CONDITIONS: Cataract; Presbyopia
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, controlled, double-masked, phased, multicenter clinical study
Who Masked: Participant, Care Provider
Masking Description: The subject will be masked to randomization assignment and will be unmasked at the completion of the study. Scheduled masked postoperative assessments will be performed by a masked examiner
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Investigational IOL (Experimental): Juvene® IOL
  Interventions: Device: Juvene IOL
- Control IOL (Active Comparator): Tecnis® Monofocal (ZCB00, PCB00 or DCB00)
  Interventions: Device: Tecnis® Monofocal (ZCB00, PCB00 or DCB00)

INTERVENTIONS:
Device: Juvene IOL — Cataract extraction and implantation of a posterior chamber IOL
  Arms: Investigational IOL
Device: Tecnis® Monofocal (ZCB00, PCB00 or DCB00) — Cataract extraction and implantation of a posterior chamber IOL
  Arms: Control IOL

SUMMARY:
To assess the safety and effectiveness of the Juvene® IOL for the treatment of aphakia and mitigation of the effects of presbyopia after removal of the natural crystalline lens due to cataract.

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects must be 22 years of age or older
* Able to comprehend and provide written informed consent
* Willing and able to comply with schedule for follow-up visits
* Demonstrate sufficient cognitive awareness to comply with examination procedures
* Other inclusion criteria specified in the protocol may apply.

Key Exclusion Criteria:

* Subjects with clinically significant dry eye syndrome (DES) expected to impact postoperative visual acuity
* Subjects taking medications that may affect ocular function (including but not limited to mydriatic, cycloplegic and miotic agents; tricyclic antidepressants, phenothiazines, benzodiazepines, first generation antihistamines, and anticholinergic agents)
* Prior intraocular or corneal surgery (including corneal refractive correction i.e., LASIK, PRK, etc.)
* Any corneal dystrophy that may affect visual acuity (e.g., keratoconus, pellucid corneal degeneration, etc.)
* Other exclusion criteria specified in the protocol may apply.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Distance-corrected intermediate ETDRS LogMar visual acuity | 12 Months
  Monocular photopic distance-corrected intermediate visual acuity (DCIVA) at 66 cm
Distance-corrected intermediate ETDRS LogMar visual acuity vs Control | 12 Months
  Monocular photopic distance-corrected intermediate visual acuity (DCIVA) statistical superiority over the Control group
Defocus curve testing with ETDRS chart | 12 Months
  Monocular diopters of depth of focus (DOF)
Best corrected distance ETDRS LogMar visual acuity vs control | 12 Months
  Monocular photopic best corrected distance visual acuity (BCDVA) statistical non-inferiority to the Control group
Best corrected distance ETDRS LogMar visual acuity | 12 Months
  Monocular photopic best corrected distance visual acuity (BCDVA)

SECONDARY OUTCOMES:
Distance-corrected near ETDRS LogMar visual acuity | 12 Months
  Monocular photopic distance-corrected near visual acuity (DCNVA) at 40 cm
Distance-corrected near ETDRS LogMar visual acuity vs control | 12 Months
  Monocular photopic distance-corrected near visual acuity (DCNVA) at 40 cm statistical superiority over the Control group

CONTACTS AND LOCATIONS:
Overall Officials: Patrick R Casey, O.D., Study Director — LensGen, Inc.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garg S, De Jesus MT, Fletcher LM, Chayet A, Barragan E, Casey P. Twelve-month clinical outcomes after implantation of a new, modular, anterior shape-changing fluid optic intraocular lens. J Cataract Refract Surg. 2022 Oct 1;48(10):1134-1140. doi: 10.1097/j.jcrs.0000000000000935. PMID 35297798
- See also: Company website — http://lensgen.com